CLINICAL TRIAL: NCT06033898
Title: Effect of the Physical Inactivity Duration on Postprandial Lipid Metabolism the Morning After Exercise
Brief Title: Inactivity Duration on Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004856
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12-hr trial (Experimental): Participants will go through a 48-hr physical activity control phase with 10,000 steps taken every 24 hours (9 pm to 9 pm the next day). This phase will be followed with a 12-hour physical inactive phase (9 pm to 9 am the next morning). Less than 1,000 steps during this 12 hours (mostly night time) will be required. The 1-hr cycling session will take place from 8 pm to 9 pm the same day when inactive phase starts. A high fat tolerance test that lasts 5 hours will take place at 9 am the last day.
  Interventions: Behavioral: 12 hours of physical inactivity
- 24-hr trial (Experimental): Participants will go through a 48-hr physical activity control phase with 10,000 steps taken every 24 hours (9 am to 9 am the next morning). This phase will be followed with a 24-hour physical inactive phase (9 am to 9 am the next morning). During this 24 hours, from 9 am to 9 pm (mostly daytime), less than 1,500 steps is required, and from 9 pm to 9 am the next morning (mostly night), less than 1,000 steps is required. The 1-hr cycling session will take place from 8 pm to 9 pm on the day when inactive phase starts. A high fat tolerance test that lasts 5 hours will take place at 9 am the last day.
  Interventions: Behavioral: 24 hours of physical inactivity
- 36-hr trial (Experimental): Participants will go through a 48-hr physical activity control phase with 10,000 steps taken every 24 hours (9 pm to 9 pm the next day). This phase will be followed with a 36-hour physical inactive phase (9 pm - 9 am on the high fat tolerance day). During the inactive phase, it includes two 12 hours that mostly at night (9 pm - 9 am the next day) and one 12 hours (9 am to 9 pm the same day) that mostly in the day. Less than 1,500 steps is required for 9 pm - 9 am periods, and less than 1,000 steps is needed for 9 am - 9 pm (same day) phase. The 1-hr cycling session will take place from 8 pm to 9 pm the second last day in the trial. A high fat tolerance test that lasts 5 hours will take place at 9 am the last day.
  Interventions: Behavioral: 36 hours of physical inactivity

INTERVENTIONS:
Behavioral: 12 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 10,000 steps per 24 hours for 48 hours, and then limit their steps below 1000 steps. A diet record form, a sleep record, and a step record form will be given to participants to log in their diet, sleep time and steps taken through out the whole trial. Participant will be asks to mimic the diet between trials.
  Arms: 12-hr trial
Behavioral: 24 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 10,000 steps per 24 hours for 48 hours, and then limit their steps below 1,000 - 1,500 steps per 12 hours for 24 hours. A diet record form, a sleep record, and a step record form will be given to participants to log in their diet, sleep time and steps taken through out the whole trial. Participant will be asks to mimic the diet between trials.
  Arms: 24-hr trial
Behavioral: 36 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 10,000 steps per 24 hours for 48 hours, and then limit their steps below 1,000 - 1,500 steps per 12 hours for 36 hours. A diet record form, a sleep record, and a step record form will be given to participants to log in their diet, sleep time and steps taken through out the whole trial. Participant will be asks to mimic the diet between trials.
  Arms: 36-hr trial

SUMMARY:
The purpose of the study is to investigate the effect of different periods of physical inactivity on postprandial lipid metabolism in the morning after exercise by measuring plasma triglyceride levels and fat oxidation (burning). The study is a crossover intervention with all healthy participants performing three trials varying in length of physical inactive (12 hours, 24 hours, and 36 hours). All trials include a physical activity control phase (>10,000 steps/24hr), a physical inactive phase (<1,000 - 1,500 steps/12hr), a moderate intensity cycling session, and a high-fat tolerance test.

DETAILED DESCRIPTION:
Physical inactivity impairs health, including contributing to chronic diseases and increasing the risk of mortality, especially related to cardiovascular diseases. Regular exercise can help reduce the risk of cardiovascular diseases, but it is not enough on its own. Prolonged sitting and having too little of light intensity of physical activity (like stepping) means lacking physical activity and is harmful for health, even for those who meet the exercise guidelines. Although an acute bout of exercise is able to improve the postprandial lipid metabolism (i.e., attenuate postprandial lipemia), it has been found that this benefit is abolished after a period of physical inactivity. Specifically, taking 8,500 steps per day or more (i.e., being physical active) would assure the benefits in postprandial lipid metabolism from exercise, while taking 5,000 steps or less (i.e., being physical inactive) would abolish this benefit from exercise. Investigators termed this phenomenon 'exercise resistance'. However, it is still unknown of how long of the of a period of physical inactive will cause 'exercise resistance'. Therefore, investigators propose this study to focuses on the effect of the length of physical inactivity on postprandial lipid metabolism the following morning after exercise. Three intervention trials differentiate with different periods of physical inactivity (12 hours, 24 hours, and 36 hours) will be involved for this purpose. The study aims to determine how long a period of physical inactivity is required for 'exercise resistance' to occur.

Twelve male and female participants will be recruited from Austin community to participate this study. All participants will self-report that they have been medically cleared for exercise by submitting a health history questionnaire. Researchers will screen all forms filled out by participants and confirm that participants are eligible for this study. Participants will receive both written and verbal descriptions of the study procedures and measurements, and provide written informed consent.

The study requires at least 7 visits besides the day for questionnaire filling and informed consent signing. One for preliminary test, and 6 for the three trials (one cycling session and one high fat tolerance tests for each trial). All visits will take place in the Human Performance Lab (BEL 820) at the University of Texas at Austin. All participants will complete one preliminary test (incremental exercise test) on a cycle ergometer before three intervention trials in a randomized order.

During the incremental exercise test, participant will cycling on a cycle ergometer with a mask. Participant's breathing air will go through the tubes connecting with the mask. By analyzing the exhaled gas during the test, the maximal oxygen consumption (VO2max) will be measured for determining the cycling intensity for the cycling in the three trials. Between trials, there will be a washout period of at least five days. The three trials varies in length of physical inactive (12 hours, 24 hours, and 36 hours). Thus, the three trials are marked as 12-hr trial, 24-hr trial, and 36-hr trial. During the cycling sessions, participant will cycle for 1 hour at an intensity of 60-65% of VO2max (moderate intensity) on a cycling ergometer. The high fat tolerance test (HFTT) day will be the day for collecting primary data.

To highlight the effect of physical inactivity duration on causing exercise resistance, all HFTT will start at the same time on the testing day of each trial, which is 9 am on the final day of each trial. For easier understanding, the events sequence in each of the trails is listed below in a backward order,

* A HFTT from 9 am to 2 pm on the last day of each trial.
* A physical inactivity phase (<1,000 - 1,500 steps/12 hr) that lasts until the beginning of the HFTT (i.e., 9 am on the last day of the trial). The lengths of this phase will be 12 hours, 24 hours, or 36 hours depending on the trial.
* A 1-hr cycling session finishing 12 hours before the HFTT (i.e., 8pm - 9pm on the second last day).
* A 48 hours of physical activity control phase (> 10,000 steps/24hr) that lasts until the beginning of the physical inactivity phase.

During the whole trials, participants will be given a pedometer for self-monitoring the step counts. A step recording form, a sleep recording form, and a diet form will be provided to participants in all trials and will be returned after each trial. A standard frozen meal will be provided to the participants to consume 2 hours before the cycling sessions to avoid the effect from fat consumption from the meal before the HFTT. Other than the sport drink that will be provided right after the cycling, participants will need to stay fasted (no food or beverage, only water) since the frozen meal to the HFTT. During the HFTT, a high fat meal (a mixture of ice cream and heavy cream) will be provided to participants. Participants will consume the milkshake in 10 min. The amount of ice cream and heavy cream will be determined by participant's body weight. During the test, five measurements (fingertip blood collection and exhaled air collection) will be done including one baseline measurement (before high fat meal), and four measurements each hour after consuming the meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between the age of 18-65 years old
* Untrained or recreationally active
* No metabolic disease, no lactose intolerance, not taking medicines altering lipid or carbohydrate metabolism
* No injury or disease affecting the cycling ability.

Exclusion Criteria:

* On medications that alter lipid or carbohydrate metabolism
* lactose intolerant
* General health problems: Heart problems or coronary artery disease, hypertension, lung or respiratory problems.
* Exercise problems: Chest pain, fainting, palpitations, told to give up sports because of health problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
Fat oxidation (fat burning) | A total of 5 measurements will be done, specifically are before the high fat meal (baseline) and each hour after the high fat meal for 4 hours. The whole test takes about 5 hours from 9 am to 2 pm on the last day of each trial.
  Exhaled gas will be collected during the high fat tolerance test. Fat oxidation will be calculated based on the gas volume and CO2 and O2 proportion.
Plasma triglyceride | A total of 5 measurements will be done, specifically are before the high fat meal (baseline) and each hour after the high fat meal for 4 hours. The whole test takes about 5 hours from 9 am to 2 pm on the last day of each trial.
  Fingertip blood will be collected during the high fat tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Jieting Wang, M.S., Principal Investigator — The University of Texas of Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No